CLINICAL TRIAL: NCT04829123
Title: A Phase 1, Double Blind, Placebo Controlled, Single and Multiple Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of HEC88473 in Healthy Subjects
Brief Title: The Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of HEC88473 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongguan HEC Biopharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC88473-DM-102
Record Dates: First submitted 2021-03-25; First posted 2021-04-02 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Single dose of 0.5 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 0.5 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 1.7 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 1.7 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 5.1 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 5.1 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 10.2 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 10.2 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 17.0 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 17.0 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 25.5 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 25.5 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 34.0 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 34.0 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Single dose of 44.2 mg HEC88473 (Experimental): Healthy subjects, receiving a single dose of 44.2 mg HEC88473 (N=6) or placebo(N=2) after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 1.7 mg HEC88473 (Experimental): Healthy subjects, receiving a weekly dose of 1.7 mg HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 5.1 mg HEC88473 (Experimental): Healthy subjects, receiving a weekly dose of 5.1 mg HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo
- Multiple doses of 10.2 mg HEC88473 (Experimental): Healthy subjects, receiving a weekly dose of 10.2 mg HEC88473 (N=10) or placebo (N=2) for 5 consecutive weeks after meal.
  Interventions: Drug: HEC88473 injection; Drug: Placebo

INTERVENTIONS:
Drug: HEC88473 injection — HEC88473 will be provided as a 17 mg/mL solution and will be administered by subcutaneous injection in the abdomen
Drug: Placebo — Placebo will be administered by subcutaneous injection in the abdomen

SUMMARY:
A Phase 1, double blind, placebo controlled, single and multiple ascending dose, safety, tolerability, pharmacokinetic, and pharmacodynamic study of HEC88473 in healthy subjects

DETAILED DESCRIPTION:
This is the first time HEC88473 will be administered to humans. The aim of this study is to obtain safety, tolerability, PK, PD, and immunogenicity data of HEC88473 SC administration as single and multiple ascending doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 60 years of age, inclusive, at screening.
2. Body weight ≥ 50 kg, and body mass index between 18.0 and 40.0 kg/m2, inclusive, at screening.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations at screening as assessed by the investigator (or designee).
4. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
3. History of alcoholism or drug/chemical abuse within 2 years prior to the first dosing.
4. Alcohol consumption of > 21 units per week for males and > 14 units per week for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
5. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at screening and/or check-in.
6. Immunization with a live attenuated vaccine or coronavirus vaccination within 1 month prior to the first dosing or planned vaccination during the course of the study.
7. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known), whichever is longer, prior to the first dosing.
8. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to first dosing, unless deemed acceptable by the investigator (or designee).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) after a single dose of HEC88473 | Baseline to day 15
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) after multiple dose of HEC88473 | Baseline to day 43
Cmax | Predose and postdose 4, 8, 10, 12, 14, 24, 48, 72, 96, 168, 216, and 336 hours
  Maximum observed plasma concentration of HEC88473
AUC | Predose and postdose 4, 8, 10, 12, 14, 24, 48, 72, 96, 168, 216, and 336 hours
  Area under the plasma concentration-time curve (AUC)

SECONDARY OUTCOMES:
OGTT | Predose and postdose 2, 4 hours
  Oral glucose tolerance test
Assessment of the incidence of anti drug antibodies (ADA) developed against HEC88473 after dosing | Baseline to day 43

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lemech, Doctor, Principal Investigator — Scientia Clinical Research
Locations (1):
- Scientia Clinical Research, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No